CLINICAL TRIAL: NCT05190432
Title: A Pilot Study of Dietary Taxifolin/Dihydroquercetin and Ergothioneine and Immune Biomarkers in Healthy Volunteers
Brief Title: Taxifolin/ergothioneine and Immune Biomarkers in Healthy Volunteers (TaxEr)
Acronym: TaxEr
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Blue California (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ERGO61222.A1
Record Dates: First submitted 2020-12-22; First posted 2022-01-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-05

CONDITIONS: Antioxidative Stress; Cold; Influenza; Aging; Inflammation
Keywords: Phagocytosis; Immunosenecence; Cytokine; Antioxidant; Metabolome; Microbiome
MeSH Terms: conditions — Common Cold; Influenza, Human; Inflammation | interventions — taxifolin; Ergothioneine

STUDY DESIGN:
Intervention Model Description: A n=90 study (3 treatment arms, each n=30) providing participants with either 250mg/day Taxifolin/DHQ, 80mg/day Ergothioneine, or control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Alphabetically labelled treatments, with de-blinding envelope held by an independent researcher at the University of Southampton.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Taxifolin/Dihydroquercetin (Experimental): 250mg/day Taxifolin (also known as Dihydroquercetin). One capsule in the morning for 8 weeks.
  Interventions: Dietary Supplement: Taxifolin
- Ergothioneine (Experimental): 80mg/day Ergothioneine. One capsule in the morning for 8 weeks.
  Interventions: Dietary Supplement: Ergothioneine
- Control (Placebo Comparator): One capsule in the morning for 8 weeks.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Taxifolin — A naturally occurring polyphenol found in apples, onions and other fruits and bark extracts.
  Other Names: Dihydroquercetin
  Arms: Taxifolin/Dihydroquercetin
Dietary Supplement: Ergothioneine — An amino acid found in mushrooms, oats and some bean varieties.
  Arms: Ergothioneine
Dietary Supplement: Control — Microcrystalline cellulose.
  Arms: Control

SUMMARY:
The complexities of the immune system make measuring the impact of dietary interventions upon its function challenging. The immune system is highly responsive to environmental influences, including the diet. An individual's diet provides the energy required to mount a strong and protective immune response, the building blocks required for synthesis of immune mediators such as antibodies and cytokines, and can also indirectly affect immune function via changes in the gut microbiome. Immune function varies across the lifecourse, with a well understood decline in immune function with age, resulting in impaired vaccination responses and an increased risk of infections and of severe complications and mortality arising from common communicable diseases such as influenza. This impaired immunity with ageing is known as immunosenescence and this affects both innate and acquired arms of the immune system.

DETAILED DESCRIPTION:
Expert guidance is available to inform the design of human nutrition trials to ensure they include the most relevant immunological outcomes (Albers, 2013). In this study, ex vivo phagocytosis and oxidative burst of immune cells will be the primary outcome, supported by other ex vivo immune measures of high clinical relevance including functional assessment of cytokine production and expression of activation markers.

Human nutritional trials frequently omit to monitor the degree of immunosenescence in participants, even amongst studies conducted amongst older adults. For example, a recent review of pre- and probiotic trials which assessed immune responses in older adults identified that only two of thirty-six studies assessed any marker of immunosenescence (Childs & Calder, 2017).

Taxifolin/DHQ is a naturally occurring polyphenol found in apples, onions and other fruits and bark extracts. Ergothioneine is an amino acid found in mushrooms, oats and some bean varieties. We hypothesise that Taxifolin/DHQ and/or Ergothioneine will alter immune function via their established antioxidant effects, and that the effects observed will vary between older adults relative to their degree of immunosenescence.

Though current dietary guidelines advise consumption of 5 portions of fruits and vegetables per day, recent surveys reveal that fewer than 30% of adults achieve this. Antioxidants found within fruits and vegetables are understood to be one of the important aspects by which our diet can influence health. It is important to investigate the effects of such antioxidants through well designed and conducted human trials.

ELIGIBILITY:
Inclusion Criteria:

* age 50-65yr
* BMI 18.5-30kg/m2
* Willing to avoid consumption of foods rich in Taxifolin/DHQ and Ergothioneine during the study period
* Willing to avoid taking any other food supplements or high doses of vitamins during the study period
* Able to provide written informed consent.

Exclusion Criteria:

* Use of prescription medication which may influence immune function, such as anti-inflammatory or immunosuppressant medication
* Diabetes requiring any medication
* Liver cirrhosis
* A history of drug or alcohol misuse
* Asplenia or other acquired or congenital immunodeficiencies
* Any autoimmune disease including connective tissue diseases
* Malignancy
* Laboratory confirmed SARS-CoV-2 infection within last 3 months
* self-reported symptoms of acute or recent infection (including use of antibiotics within the last 3 months)

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Phagocytosis activity by granulocytes ex vivo | 8 weeks post intervention
  Mean fluorescence intensity per cell will be assessed by flow cytometry.

SECONDARY OUTCOMES:
Percentage phagocytosis by monocytes ex vivo | 4 weeks, 8 weeks, 3 months post intervention
  Percentage of cells undergoing phagocytosis will be assessed by flow cytometry.
Phagocytosis activity by monocytes ex vivo | 4 weeks, 8 weeks, 3 months post intervention
  Mean fluorescence intensity per cell will be assessed by flow cytometry.
Percentage phagocytosis by granulocytes ex vivo | 4 weeks, 8 weeks, 3 months post intervention
  Percentage of cells undergoing phagocytosis will be assessed by flow cytometry.
Phagocytosis activity by granulocytes ex vivo | 4 weeks, 3 months post intervention
  Mean fluorescence intensity per cell will be assessed by flow cytometry.
Percentage oxidative burst by monocytes ex vivo | 4 weeks, 8 weeks, 3 months post intervention
  Percentage of cells undergoing oxidative burst will be assessed by flow cytometry.
Oxidative burst activity by monocytes ex vivo | 4 weeks, 8 weeks, 3 months post intervention
  Mean fluorescence intensity per cell will be assessed by flow cytometry.
Percentage oxidative burst by granulocytes ex vivo | 4 weeks, 8 weeks, 3 months post intervention
  Percentage of cells undergoing oxidative burst will be assessed by flow cytometry.
Oxidative burst activity by granulocytes ex vivo | 4 weeks, 8 weeks, 3 months post intervention
  Mean fluorescence intensity per cell will be assessed by flow cytometry.
Frequencies of naive T cells | 8 weeks
  The proportion of naive T cells will be assessed by flow cytometry.
Frequencies of memory T cells | 8 weeks
  The proportion of memory T cells will be assessed by flow cytometry.
CD57 expression upon T cells. | 8 weeks
  The proportion of T cells expressing CD57 (a marker associated with chronic immune activation) and the mean fluorescence intensity per cell will be assessed by flow cytometry.
CD28 expression upon T cells. | 8 weeks
  The proportion of T cells expressing CD28 (a cell surface marker required for T cell activation and survival) and the mean fluorescence intensity per cell will be assessed by flow cytometry.
Plasma lipid peroxides | 8 weeks
  Participant plasma lipid peroxides will be measured by colorimetric analysis.
Urinary isoprostanes | 4 weeks, 8 weeks, 3 months post intervention
  Participant urinary isoprostanes will be measured by commercially available ELISA.
Plasma isoprostanes | 4 weeks, 8 weeks, 3 months post intervention
  Participant plasma isoprostanes will be measured by commercially available ELISA.
Cytokine production by cryopreserved peripheral blood mononuclear cells in response to lipopolyssaccharide | 4 weeks, 8 weeks
  A panel of pro- and anti-inflammatory cytokines secreted by immune cells ex vivo will be assessed by Luminex array.
Cytokine production by cryopreserved peripheral blood mononuclear cells in response to influenza or coronavirus vaccine products | 4 weeks, 8 weeks
  A panel of pro- and anti-inflammatory cytokines secreted by immune cells ex vivo will be assessed by Luminex array.
Metabolomic analysis of urine samples | 4 weeks, 8 weeks, 3 months post intervention
  Full metabolic profiling of first-morning urine samples will be used to assess changes to metabolic activity of participants and their microbiome.
Metabolomic analysis of serum samples | 4 weeks, 8 weeks, 3 months post intervention
  Full metabolic profiling of serum samples will be used to assess changes to metabolic activity of participants.
Faecal microbiome analysis | 4 weeks, 8 weeks, 3 months post intervention
  Sequences of ribosomal RNA (rRNA) in participant faecal samples will be measured to assess changes in the numbers or proportions of bacterial genera and species/strains.
Incidence of self-reported seasonal cold, coronavirus and influenza-like illness. | 4 weeks, 8 weeks, 3 months post intervention
  A daily online form will be completed by participants to log any seasonal cold, coronavirus and influenza-like illness.
Duration of self-reported illness. | 4 weeks, 8 weeks, 3 months post intervention
  A daily online form will be completed by participants to log any self-reported illness.
Severity of self-reported illness. | 4 weeks, 8 weeks, 3 months post intervention
  A daily online form will be completed by participants to log any self-reported illness.
Self-reported medication use. | 4 weeks, 8 weeks, 3 months post intervention
  A daily online form will be completed by participants to log any medication use.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline E Childs, PhD, Principal Investigator — University of Southampton
Locations (1):
- NIHR Southampton Biomedical Research Centre, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albers R, Bourdet-Sicard R, Braun D, Calder PC, Herz U, Lambert C, Lenoir-Wijnkoop I, Meheust A, Ouwehand A, Phothirath P, Sako T, Salminen S, Siemensma A, van Loveren H, Sack U. Monitoring immune modulation by nutrition in the general population: identifying and substantiating effects on human health. Br J Nutr. 2013 Aug;110 Suppl 2:S1-30. doi: 10.1017/S0007114513001505. PMID 23902657
- [Background] Childs, C. E., & Calder, P. C. (2017). Modifying the gut microbiome through diet: effects on the immune system of elderly subjects. In T. Fulop, C. Franceschi, K. Hirokawa, & G. Pawelec (Eds.), Handbook of Immunosenescence Cham: Springer International Publishing AG. DOI: 10.1007/978-3-319-64597-1_160-1
- [Background] EFSA Panel on Dietetic Products, Nutrition and Allergies (NDA); Turck D, Bresson JL, Burlingame B, Dean T, Fairweather-Tait S, Heinonen M, Hirsch-Ernst KI, Mangelsdorf I, McArdle HJ, Naska A, Neuhauser-Berthold M, Nowicka G, Pentieva K, Sanz Y, Siani A, Sjodin A, Stern M, Tome D, Vinceti M, Willatts P, Engel KH, Marchelli R, Poting A, Poulsen M, Schlatter J, Gelbmann W, Van Loveren H. Scientific Opinion on taxifolin-rich extract from Dahurian Larch (Larix gmelinii). EFSA J. 2017 Feb 14;15(2):e04682. doi: 10.2903/j.efsa.2017.4682. eCollection 2017 Feb. PMID 32625400
- [Background] EFSA Panel on Dietetic Products, Nutrition and Allergies (NDA); Turck D, Bresson JL, Burlingame B, Dean T, Fairweather-Tait S, Heinonen M, Hirsch-Ernst KI, Mangelsdorf I, McArdle HJ, Naska A, Neuhauser-Berthold M, Nowicka G, Pentieva K, Sanz Y, Siani A, Sjodin A, Stern M, Tome D, Vinceti M, Willatts P, Engel KH, Marchelli R, Poting A, Poulsen M, Schlatter JR, Ackerl R, van Loveren H. Statement on the safety of synthetic l-ergothioneine as a novel food - supplementary dietary exposure and safety assessment for infants and young children, pregnant and breastfeeding women. EFSA J. 2017 Nov 13;15(11):e05060. doi: 10.2903/j.efsa.2017.5060. eCollection 2017 Nov. PMID 32625352
- [Background] Vega-Villa KR, Remsberg CM, Ohgami Y, Yanez JA, Takemoto JK, Andrews PK, Davies NM. Stereospecific high-performance liquid chromatography of taxifolin, applications in pharmacokinetics, and determination in tu fu ling (Rhizoma smilacis glabrae) and apple (Malus x domestica). Biomed Chromatogr. 2009 Jun;23(6):638-46. doi: 10.1002/bmc.1165. PMID 19267323
- [Background] Ey J, Schomig E, Taubert D. Dietary sources and antioxidant effects of ergothioneine. J Agric Food Chem. 2007 Aug 8;55(16):6466-74. doi: 10.1021/jf071328f. Epub 2007 Jul 6. PMID 17616140
- [Background] Przemska-Kosicka A, Childs CE, Enani S, Maidens C, Dong H, Dayel IB, Tuohy K, Todd S, Gosney MA, Yaqoob P. Effect of a synbiotic on the response to seasonal influenza vaccination is strongly influenced by degree of immunosenescence. Immun Ageing. 2016 Mar 15;13:6. doi: 10.1186/s12979-016-0061-4. eCollection 2016. PMID 26985232
- [Background] Ohara O. [Rapid cDNA sequencing method using the polymerase chain reaction]. Tanpakushitsu Kakusan Koso. 1990 Oct;35(14):2319-28. No abstract available. Japanese. PMID 2267325
- [Background] Taves DR. Minimization: a new method of assigning patients to treatment and control groups. Clin Pharmacol Ther. 1974 May;15(5):443-53. doi: 10.1002/cpt1974155443. No abstract available. PMID 4597226